CLINICAL TRIAL: NCT04316195
Title: Electromyographic Evaluation of the Bulbocavernosus Reflex After Acute Spinal Cord Injury: a New Prognostic Concept
Brief Title: Evaluation of the Bulbocavernosus Reflex After Acute Spinal Cord Injury
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Andréane Richard-Denis (Other)
Responsible Party: Sponsor-Investigator, Andréane Richard-Denis, MD. MSc. Physiatrist in Physical Medicine and Rehabilitation following spinal cord injury, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Organization: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Other Study IDs: 2019-1709
Record Dates: First submitted 2020-03-18; First posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Bulbocavernosus Reflex; Spinal Cord Injuries
Keywords: Bulbocavernosus reflex following a traumatic spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient admitted for an acute traumatic spinal cord injury
  Interventions: Diagnostic Test: Assessment of the bulbocavernosus reflex

INTERVENTIONS:
Diagnostic Test: Assessment of the bulbocavernosus reflex — According to the International Standards for Neurological Classification of Spinal Cord : The standard examination consists of the contraction of the bulbocavernous muscle following stimulation of the glans of the penis in men and of the clitoris in women.
  By electromyography: The electromyography consists to stimulate the bulbocavernosus reflex with a bipolar probe apply on the glans for men, and on the clitoris in women. A surface electrode will be positioned on the right or left bulbocavernous muscle at the base of the penis (or vagina) and the anus for recording. The bulbocavernous reflex will be obtained by stimulation at a frequency of 1.5Hz and an amplitude of 14 to 47 mA.

SUMMARY:
The purpose of this study is to evaluate the possibility to use electromyography in acute phase after a traumatic spinal cord injury to measure quantitatively and objectively the bulbocavernosus reflex. This study also aims to determine if there is a relationship between the bulbocavernosus reflex and neuro-functional recovery 3 months after a traumatic spinal cord injury. To do so, 20 patients admitted for acute traumatic spinal cord injury will be recruited prospectively. Within 72 hours post-trauma, the bulbocavernous reflex of all participants will be assessed according to the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) and by electromyography. Neurological improvement during the rehabilitation process and functional status at 3 months following the traumatic spinal cord injury will also be assessed.

DETAILED DESCRIPTION:
Traumatic spinal cord injuries cause severe neurological deficits (motor, sensory and autonomic disorders). Affected individuals have functional limitations and a reduced quality of life that result in high medical and social costs. Some studies have shown that early rehabilitation improves recovery. It seems therefore essential to optimize patient management in the acute phase in order to improve interventions and optimize their functional recovery.

A major barrier to early patient management is associated with a lack of knowledge about the neurophysiological mechanisms of acute spinal cord injury. Moreover, early assessment of prognosis is still difficult to make. The early assessment is based almost exclusively on the clinical neurological examination and does not include an objective measurement of underlying neurophysiological processes. The possibility to establish an accurate neuro-functional prognosis at an early stage will have the advantage to guide clinical decision, allow the development of an appropriate rehabilitation plan and figure out the long-term needs of the patient while promoting better collaboration.

Clinical neurological examination includes among other things, the evaluation of the bulbocavernosus reflex. The purpose of this study is to evaluate the possibility to use electromyography in acute phase after a traumatic spinal cord injury to measure quantitatively and objectively the bulbocavernosus reflex. This study also aims to determine if there is a relationship between the bulbocavernous reflex and neuro-functional recovery 3 months after a traumatic spinal cord injury.

The bulbocavernous reflex of patients admitted for acute traumatic spinal cord injury will be assessed within 72 hours post-trauma according to the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) and by electromyography. Neurological improvement during the rehabilitation process and functional status at 3 months following the traumatic spinal cord injury will also be assessed. Descriptive analyses will be proposed to characterize the bulbocavernous reflex obtained by electromyography evaluation. Comparative analyses will be carried out to describe the characteristics of patients with different bulbocavernosus reflex stimulation thresholds. Correlations will also be established to determine the relationship between the electromyography evaluation of the bulbocavernosus reflex and the neurological and functional improvement of the patient.

ELIGIBILITY:
Inclusion Criteria:

* male or female age of 18 years or older
* patient with fracture, fracture-dislocation or vertebral dislocation from C0 to T12 inclusively
* patient with neurological impairment involving the motor spinal cord (severity AIS grade A or B) on initial assessment
* patient admitted to Hôpital du Sacré-Coeur de Montréal within 72 hours for trauma
* patient transfer to intensive functional rehabilitation

Exclusion Criteria:

* pregnancy
* suspicion of sacral nerve damage (caused by trauma or other co-morbidities)
* spinal cord syndrome (caused by trauma or other comorbidities) or spinal cord signal abnormality on magnetic resonance imaging
* pre-existing major neurological impairment (e.g. stroke, Parkinson's disease, etc.)
* inability to consent (coma, delirium, etc.)
* perineal injury preventing the sacral EMG procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient admitted to the Hôpital du Sacré-Coeur de Montréal for a traumatic spinal injury.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Characterize the bulbocavernosus reflex using electromyographic assessment within 72 hours of a traumatic spinal cord injury | During the acute care hospitalization, max 72 hours
  Determine stimulation threshold, latency and amplitude of the signal
Determine the relationship between the bulbocavernosus reflex and the neurological and functional recovery of patients 3 months after a traumatic spinal cord injury | After hospitalization, 3 months post operation
  Related neurological and functional improvement according to acute electromyographic reflex measurement

CONTACTS AND LOCATIONS:
Overall Officials: Andréane Richard-Denis, M.D., MSC., Principal Investigator — CIUSSS du Nord-de-l'Île-de-Montréal-Hôpital du Sacré-Cœur de Montréal
Locations (1):
- CIUSSS du Nord-de-l'île-de-Montréal-Hôpital du Sacré-Cœur de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Richard-Denis A, Beausejour M, Thompson C, Nguyen BH, Mac-Thiong JM. Early Predictors of Global Functional Outcome after Traumatic Spinal Cord Injury: A Systematic Review. J Neurotrauma. 2018 Aug 1;35(15):1705-1725. doi: 10.1089/neu.2017.5403. Epub 2018 Apr 17. PMID 29455634
- [Background] Simpson LA, Eng JJ, Hsieh JT, Wolfe DL; Spinal Cord Injury Rehabilitation Evidence Scire Research Team. The health and life priorities of individuals with spinal cord injury: a systematic review. J Neurotrauma. 2012 May 20;29(8):1548-55. doi: 10.1089/neu.2011.2226. Epub 2012 Apr 18. PMID 22320160
- [Background] Richard-Denis A, Thompson C, Mac-Thiong JM. Quality of life in the subacute period following a cervical traumatic spinal cord injury based on the initial severity of the injury: a prospective cohort study. Spinal Cord. 2018 Nov;56(11):1042-1050. doi: 10.1038/s41393-018-0178-8. Epub 2018 Jul 3. PMID 29970920
- [Background] Krueger H, Noonan VK, Trenaman LM, Joshi P, Rivers CS. The economic burden of traumatic spinal cord injury in Canada. Chronic Dis Inj Can. 2013 Jun;33(3):113-22. English, French. PMID 23735450
- [Background] Hachem LD, Ahuja CS, Fehlings MG. Assessment and management of acute spinal cord injury: From point of injury to rehabilitation. J Spinal Cord Med. 2017 Nov;40(6):665-675. doi: 10.1080/10790268.2017.1329076. Epub 2017 Jun 1. PMID 28571527
- [Background] Dvorak MF, Noonan VK, Fallah N, Fisher CG, Rivers CS, Ahn H, Tsai EC, Linassi AG, Christie SD, Attabib N, Hurlbert RJ, Fourney DR, Johnson MG, Fehlings MG, Drew B, Bailey CS, Paquet J, Parent S, Townson A, Ho C, Craven BC, Gagnon D, Tsui D, Fox R, Mac-Thiong JM, Kwon BK. Minimizing errors in acute traumatic spinal cord injury trials by acknowledging the heterogeneity of spinal cord anatomy and injury severity: an observational Canadian cohort analysis. J Neurotrauma. 2014 Sep 15;31(18):1540-7. doi: 10.1089/neu.2013.3278. Epub 2014 Jul 8. PMID 24811484
- [Background] Kirshblum SC, Burns SP, Biering-Sorensen F, Donovan W, Graves DE, Jha A, Johansen M, Jones L, Krassioukov A, Mulcahey MJ, Schmidt-Read M, Waring W. International standards for neurological classification of spinal cord injury (revised 2011). J Spinal Cord Med. 2011 Nov;34(6):535-46. doi: 10.1179/204577211X13207446293695. No abstract available. PMID 22330108
- [Background] Consortium for Spinal Cord Medicine. Early acute management in adults with spinal cord injury: a clinical practice guideline for health-care professionals. J Spinal Cord Med. 2008;31(4):403-79. doi: 10.1043/1079-0268-31.4.408. No abstract available. PMID 18959359
- [Background] Podnar S. Neurophysiologic studies of the penilo-cavernosus reflex: normative data. Neurourol Urodyn. 2007;26(6):864-9. doi: 10.1002/nau.20411. PMID 17335052
- [Background] Granata G, Padua L, Rossi F, De Franco P, Coraci D, Rossi V. Electrophysiological study of the bulbocavernosus reflex: normative data. Funct Neurol. 2013 Oct-Dec;28(4):293-5. PMID 24598398
- [Background] Fehlings MG, Tetreault LA, Aarabi B, Anderson P, Arnold PM, Brodke DS, Chiba K, Dettori JR, Furlan JC, Harrop JS, Hawryluk G, Holly LT, Howley S, Jeji T, Kalsi-Ryan S, Kotter M, Kurpad S, Kwon BK, Marino RJ, Martin AR, Massicotte E, Merli G, Middleton JW, Nakashima H, Nagoshi N, Palmieri K, Singh A, Skelly AC, Tsai EC, Vaccaro A, Wilson JR, Yee A, Burns AS. A Clinical Practice Guideline for the Management of Patients With Acute Spinal Cord Injury: Recommendations on the Type and Timing of Rehabilitation. Global Spine J. 2017 Sep;7(3 Suppl):231S-238S. doi: 10.1177/2192568217701910. Epub 2017 Sep 5. PMID 29164029